CLINICAL TRIAL: NCT02599831
Title: Efficacy of Electrical Pudendal Nerve Stimulation for Patients With Post Prostatectomy Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZYSNXD-CC
Record Dates: First submitted 2015-10-29; First posted 2015-11-09 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2017-12

CONDITIONS: Urinary Incontinence
Keywords: Electrical pudendal nerve stimulation; Pelvic floor muscle training; Transanal electrical stimulation; Post radical prostatectomy incontinence; Comparative study
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrical pudendal nerve stimulation (Experimental): Four sacrococcygeal points were selected. Two 0.40Х100 mm needles were inserted perpendicularly to a depth of 80-90 mm 1 cm bilateral to the sacrococcygeal joint, to produce a sensation referred to the root of the penis (perineum) or the anus. Two needles of 0.40Х100 or 125mm were inserted obliquely toward the ischiorectal fossa to a depth of 90 to 110 mm about 1 cm bilateral to the tip of the coccyx, to produce a sensation referred to the root of the penis (or the perineum).
  Each two ipsilaterally needles were connected to one electrode from a G6805-2Multi-Purpose Health Device (Shanghai Medical Instruments High-Techno, Shanghai, China), with a frequency of 2.5 Hz and an intensity (45~55 mA). EPNS was given for 60 min a time, 3 times per week for 8 weeks.
  Interventions: Device: Electrical pudendal nerve stimulation
- PFM training with Transanal ES (Active Comparator): Electromyogram BF-assisted PFMT (using a nerve function reconstruction treatment system (AM1000B; Shenzhen Creative Industry Co. Ltd, China) and following TES (using a neuromuscular stimulation therapy system (PHENIX USB4, Electronic Concept Lignon Innovation, France)) at a current intensity of < 60 mA (as high as possible within the patient's tolerance) and frequencies of 15 Hz and 85 Hz (alternate 3-minute periods of stimulation) were performed by a specially trained therapist, 20 minutes each time, respectively (a total of 40 minutes), 3 times a week for a total of 8 weeks. The patients were also required to conduct 30 maximal high-intensity PFM contractions for 2-6 seconds (with 2-6 seconds rest), 3 sessions every day at home for a total of 8 weeks.
  Interventions: Device: PFM training; Device: Transanal ES

INTERVENTIONS:
Device: Electrical pudendal nerve stimulation — Four sacrococcygeal points are selected. The two upper points are located about 1 cm bilateral to the sacrococcygeal joint. On the upper points, a needle of 0.40 Х 100 mm is inserted perpendicularly to a depth of 80 to 90 mm to produce a sensation referred to the root of the penis (perineum) or the anus. The locations of the two lower points are about 1 cm bilateral to the tip of the coccyx. On the lower points, a needle of 0.40 Х 100 or 125 mm is inserted obliquely towards the ischiorectal fossa to a depth of 90 to 110 mm to produce a sensation referred to the root of the penis (perineum). After the sensation referred to the above regions is produced, each of two pairs of electrodes from a G6805-2 Multi-Purpose Health Device is connected with the two ipsilaterally inserted needles.
  Other Names: G6805-2 Multi-Purpose Health Device
  Arms: Electrical pudendal nerve stimulation
Device: PFM training — A nerve function reconstruction treatment system (AM1000B; Shenzhen Creative Industry Co.Ltd, China) is used for EMG-biofeedback assisted PFMT.
  Other Names: AM1000B (Shenzhen Creative Industry Co.Ltd, China)
  Arms: PFM training with Transanal ES
Device: Transanal ES — A neuromuscular stimulation therapy system (PHENIX USB 4，Electronic Concept Lignon Innovation, France) is used for TES
  Arms: PFM training with Transanal ES

SUMMARY:
The purpose of this study is to determine whether electrical pudendal nerve stimulation is more effective than pelvic floor muscle training plus transanal electrical stimulation in treating post prostatectomy Incontinence.

DETAILED DESCRIPTION:
Conservative therapy could be considered a choice of treatment for stress urinary incontinence (SUI) as it seems to have no side effect and causes significant and long-term improvement in symptoms. Pelvic floor muscle training (PFMT) and electrical stimulation are two commonly used forms of conservative treatment for SUI. PFMT improves the structural support of the pelvis. However, many patients have difficulty identifying and isolating their pelvic floor muscles (PFM) and are unable to perform the exercise effectively. Furthermore, patients who can identify the PFM often find that the required daily exercise routine is burdensome. Hence, the primary disadvantage of PFMT is lack of long-term patient compliance. Electrical stimulation (ES) is a non-invasive, passive treatment that produces a muscle contraction. Transanal electrical stimulation (TES) has little side-effect, and the patient compliance is 70-85% in published reports. TES results in PFM contraction by indirect nerve stimulation, mainly by polysynaptic reflex responses. The indirect stimulation and reflexive contraction may be the reason why the effect of electrical stimulation is not as good as that of PFMT when performed correctly. By combining the advantages of PFMT and TES and incorporating the technique of deep insertion of long acupuncture needles, we developed electrical pudendal nerve stimulation (EPNS). In EPNS, long acupuncture needles of 0.40 Х 100 or 125 mm were deeply inserted into four sacral points and electrified to stimulate the pudendal nerves (PN) and contract the PFM. CT transverse plane at the coccygeal apex has showed that the position of the lower needle tip is similar to where (adjacent to PN at Alcock's canal) the Bion device is implanted for chronic PN stimulation. Our previous study showed that EPNS had a better therapeutic effect on female SUI as compared with PFMT + TES. Simultaneous records of perineal ultrasonographic PFM contraction, vaginal pressure and pelvic floor surface electromyogram in our previous study have proved that EPNS can exactly excite PN and induce PFM contraction in female SUI patients. However, EPNS has also shown satisfactory effect in male patients with SUI problems. The purpose of this study is to compare the efficacy of EPNS to PFMT + TES in treating male SUI.

ELIGIBILITY:
Inclusion Criteria:

* incontinence at 1 month or more after RP
* ≥2 incontinence episodes a week on baseline 7-day bladder diary
* no residual cancer after RP on pathological examination

Exclusion Criteria:

* the presence of preoperative incontinence
* treatment with anticholinergics
* urinary tract infection or hematuria
* postvoid residual volume>100 mL

Ages: 25 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
ICIQ-UI-SF | 8 weeks
  International Consultation on Incontinence Questionnaire-Urinary Incontinence-Short Form

SECONDARY OUTCOMES:
diaper numbers | 8 weeks
  none, 1-3 per week, 4-6 per week, 1-4 per day and more than 4 per day are scored 0, 1, 2, 3 and 4 respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai research institute of acupuncture and meridian, Shanghai, China